CLINICAL TRIAL: NCT05437276
Title: A Therapeutic Experience Program (TEP) Study Assessing Adherence to On-Label PoNS® Therapy for Improvement of Gait in People With Multiple Sclerosis (MS) in a Real-World Clinical Setting
Brief Title: A Therapeutic Experience Program (TEP) Study for Improvement of Gait in People With Multiple Sclerosis (MS)
Acronym: PoNSTEP
Status: Completed | Type: Observational
Sponsor: Helius Medical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: HMI-MS-PoNS-TE001
Record Dates: First submitted 2022-06-17; First posted 2022-06-29 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Gait Impairment Due to Mild/Moderate Multiple Sclerosis (MS)
Keywords: Gait, rehabilitation, PoNS, device, therapy, adherence, outcome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- People with mild to moderate Multiple Sclerosis and gait deficit: All enrolled subjects will go through 14 weeks therapy: Phase 1 (2-week in-clinic supervised PoNS therapy) followed by Phase 2 (12-week period of at-home unsupervised - PoNS therapy).
  Six-Month Observation: subjects will be asked to return to the clinic six months after the end of the 14-week course of therapy for an observation visit.
  Individual subjects could receive, upon investigator's opinion of need, an ad hoc second 12-week course of PoNS therapy.
  Interventions: Device: PoNS®

INTERVENTIONS:
Device: PoNS® — The PoNS device used in conjunction with rehabilitative physical therapy

SUMMARY:
PoNS therapy is a rehabilitation program that uses the PoNS device in conjunction with individualized physical exercise. This is an outcome research open label observational interventional multi-center study investigating the relationship between subject's adherence to PoNS therapy and therapeutic outcomes.

DETAILED DESCRIPTION:
Study participants will undergo fourteen weeks of on-label PoNS therapy and, specifically, two weeks in-clinic PoNS therapy directly supervised by a physical therapist who has been trained on PoNS therapy by Helius Medical and certified as a clinic PoNS trainer (Phase 1) followed by 12 weeks of at-home unsupervised PoNS therapy Once weekly in-clinic PoNS therapy session (Phase 2). Subjects will be then asked to return to the clinic six month after the end of the study Phase 2 to assess maintenance of PoNS therapy effects.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 22 years of age with a diagnosis of MS.
2. EDSS scores < 6.5 at screening; a demonstrated gait deficit.
3. Can walk at least 10 meters with or without the use of walking aids.
4. Participants must be stable without relapse for at least 60 days and agree to PoNS therapy regimen.

Exclusion Criteria:

1. Other neurological, visual, or orthopedic problems that significantly interfere with balance or gait.
2. Dementia.
3. Subjects who are currently attending physical rehabilitation and are unwilling to switch to PoNS-specific physical therapy regimen.
4. Subjects who are already functional community ambulators (gait speed>120cm/s43).
5. Subjects will also be excluded as per the Helius Medical PoNS device indication for usage ("electrical stimulation should not be used: if there is an active or suspected malignant tumor; in areas of recent bleeding or open wounds; in areas that lack normal sensation; in women who are pregnant, or in people with sensitivity to nickel, gold or copper").

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 50 subjects across 10-12 clinical sites in the U.S. will participate in this study. Candidates with scores < 6.5 on the Kurtzke Expanded Disability Status Scale (EDSS) (from mild impairment up to use of an assistive device) will be considered for participation. Subjects will have no major co-morbidities (e.g., neurological disorders, uncontrolled pain, hypertension, or diabetes). All subjects, if on medications, will not have had any major changes in type or dosage of medication within three months of enrollment. Subjects with oral health problems or neurological disorders other than those attributed to their primary diagnosis will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Measure subjects' adherence to PoNS therapy (device + physical therapy) | 14 weeks
  Subjects' adherence to at-home PoNS therapy (device + physical therapy) over 12 weeks following 2 weeks of supervised PoNS therapy at a physical therapy clinic and the relationship between subject's therapy adherence behavior and therapeutic functional outcomes as measured by the Dynamic Gait Index (DGI).

SECONDARY OUTCOMES:
1) Clinical improvement and its relationship to adherence over the 14-week course of PoNS therapy by evaluating | 14 weeks
  a. subject's improvement of gait as measured by the Timed 25-foot Walk Test
1) Clinical improvement and its relationship to adherence over the 14-week course of PoNS therapy by evaluating | 14 weeks
  b. balance deficits as measured by the Timed Up and Go Cognitive (TUG-Cog) Test,
1) Clinical improvement and its relationship to adherence over the 14-week course of PoNS therapy by evaluating | 14 weeks
  c. investigator's impression of clinical improvement as measured by the Clinical Global Impression (CGI)
Clinical improvement among subjects receiving a second course of PoNS therapy as measured by: | 14 weeks
  a. the rate and timing of investigator initiated second course of therapy
Clinical improvement among subjects receiving a second course of PoNS therapy as measured by: | 14 weeks
  b. the magnitudes of improvements in gait and balance deficits during the second course of therapy
3) Association between likelihood of second course of therapy and magnitudes of improvement with adherence during the initial therapy | 14 weeks
  adherence during the second course of therapy, and changes in adherence

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Favit-VanPelt, Study Director — Helius Medical Inc
Locations (5):
- United States (5):
  - Shepherd Center, Atlanta, Georgia
  - MGH Institute of Health Professions, Boston, Massachusetts
  - Neurology Center of New England, P.C., Foxborough, Massachusetts
  - NYU Langone Health, NYU Grossman School of Medicine, New York, New York
  - Oregon Health and Science university (OHSU), Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
All participating investigators will have access to deidentified individual patient data
Supporting Information: Study Protocol, CSR
Time Frame: Study duration
Access Criteria: Participant investigators